CLINICAL TRIAL: NCT05638113
Title: Prolonged Air Leakage After Major Lung Resection
Acronym: PRAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Finn Ørjar Amundsen Dittberner, Principal Investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20220068
Record Dates: First submitted 2022-11-17; First posted 2022-12-06 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Air Leak
Keywords: Blood pleurodesis

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood pleurodesis (Active Comparator)
  Interventions: Procedure: Pleural injection of autologous blood
- Simple chest drainage (chest tube) (No Intervention)

INTERVENTIONS:
Procedure: Pleural injection of autologous blood — 120 ml autologous blood will be drawn from simple venous puncture and immediately injected through the drain into the pleural cavity followed by flushing with 50ml of saline.
  Arms: Blood pleurodesis

SUMMARY:
The goal of this prospective randomized controlled trial is to investigate the clinical effects of autologous blood pleurodesis in the treatment of pulmonary air leaks on the first postoperative day following VATS pulmonary resections. Patients will through web-based randomization be randomly assigned into intrapleural instillation of autologous blood (intervention) or standard treatment with ordinary chest drainage (control).

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial enrolling patients undergoing elective VATS-lobectomy. Patients will be randomly assigned into two groups through web-based randomization. Air leak will be measured intraoperatively by submersion tests and postoperatively using standard electronic chest tube devices (Thopaz) with a regulated pressure of -10 cmH2O. If an air leak is present on the 1st postoperative day (20 ml/min or greater for at least 6 hours) patients will be invited to participate in this study.

Following informed consent, the patient is randomized on a web-based randomization module to receive intervention or observation. The intervention group will receive intrapleural instillation of autologous blood in accordance with the standard blood patch protocol at Odense University Hospital. In short, 120 ml autologous blood will be drawn from simple venous puncture and immediately injected through the drain into the pleural cavity followed by flushing with 50ml of saline. No anticoagulation or coagulating agents will be added. All other aspects of the patient's postoperative management will be according to the department's standard protocols.

Standard preoperative information on smoking status, medications, medical history of lung diseases, BMI, spirometry as well as DLCO measurements will be recorded. Detailed information about the surgical treatment will also be recorded (site of anatomical resection, adherences, standard perioperative assessment of air leakage, and type of mechanical linear staplers).

All chest drains will be connected to a standard electronic chest tube device (Thopaz) for continuous recording of air leakage and the drain is removed during daytime or evening shifts when air leakage has ceased to 20 ml/min or less for at least 6 hours according to the standard postoperative management. In addition, all included patients will undergo standard postoperative observations, including recording of vital signs (blood pressure, heart rate, fever, saturation-%) and standard blood samples (CRP and leukocyte count) on postoperative day 2 and subsequent daily if there is a suspicion of infection, pleural effusions, empyema and drain-site infections. Pain will be assessed twice daily using a standardized 0-10 visual analog scale (VAS) where 0 represents no pain and 10 the worst imaginable pain.

Electronic recordings of air leakage from the electronic chest tube device will be analyzed from drain placement in the operating room, until drain removal. If air leakage is still present on postoperative day 7, treatment is considered a failure and further management will be individualized by the responsible surgeon including the need for re-operation in accordance with the department's standard of care.

In the control group everything listed above will apply in the same manner except the intrapleural instillation of autologous blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Patients willing to give informed consent
* Patients undergoing VATS lobectomy
* Patients with a postoperative air leak (> 20ml/min for at least 6 hours).

Exclusion Criteria:

* Patients < 18 years of age
* Patients not willing to give informed consent
* Trauma patients
* Hypotensive patients and patients with a low blood cell count (anemia, thrombocytopenia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Duration of air leakage until sealed. | Through study completion, an average of 3 years.
  Outcome measure will be assessed when the electronic drain box indicates no further air leak. Data will be reported as hours of air leakage until sealed.
Duration until chest drain removal. | Through study completion, an average of 3 years.
  Outcome measure will be assessed when the patients chest drain is removed. Data will be reported as hours with chest drain until removed.
Duration of hospital stay. | Through study completion, an average of 3 years.
  Outcome measure will be assessed when the patient is discharged from the hospital. Data will be reported as days hospitalized until discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Licht, Professor, Study Director — Odense University Hospital
Locations (1):
- Department of Cardiothoracic Surgery, Odense University Hospital, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No